CLINICAL TRIAL: NCT06192602
Title: Testing the Effectiveness of an Acceptance-based Adherence Therapy for People With Recent-onset Psychosis: A Randomized Controlled Trial
Brief Title: Effects of an Acceptance-based Medication Adherence Therapy for Recent-onset Psychosis
Acronym: AIM_AT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Integrated Community Centers for Mental Wellness (Unknown)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 19202171
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Early Psychosis; Psychotic Disorders
Keywords: recent-onset psychosis; randomized controlled trial; insight into illness; acceptance; psychotic symptoms; rehospitalization; medication adherence; service satisfaction
MeSH Terms: conditions — Psychotic Disorders; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Assessor-blind, repeated measures, parallel-group randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome assessors, researchers and center staff are blind to the group assignment and intervention undertaken, and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acceptance-based, insight-inducing medication adherence therapy (AIM-AT) (Experimental): Acceptance-based Insight-inducing and Medication Adherence Therapy (AIM_AT) consists of 10 weekly/biweekly, 2-hour sessions (4-months), based on the modified Kemp's model/manual of Adherence therapy and mindfulness-based psychoeducation program developed by the research team. The integrative AIM_AT program based on the principles of motivational-interviewing technique (MI) and mindfulness- and acceptance-based therapy, which have been tested in our previous controlled trials and increasingly been shown to reduce both positive and negative psychotic symptoms and ambivalent attitude towards medication adherence and inducing treatment/illness insight.
  Interventions: Behavioral: AIM_AT; Behavioral: TAU
- Conventional Psychoeducation Group program (CPG) (Active Comparator): Psychoeducation groups (12-18 members/group) will be led by one trained psychiatric nurse in each center experienced in psychiatric rehabilitation, and are guided by a validated group-intervention protocol based on the research team's and McFarlane et al.'s psychoeducation programs for psychosis. The psychoeducation program consists of 10 two-hour sessions, weekly/biweekly (similarly, 4-month duration) and is comprised of six components: introduction and goal-setting; basic understanding of psychosis and symptom and emotion self-care; education workshop of psychosis care, treatment and community support services; learning about self-care skills; establishing social support and effective coping skills; and skills practices, review and future plan.
  Interventions: Behavioral: CPG; Behavioral: TAU
- Treatment-as-usual only (TAU) (Other): Routine/Usual care only (control) group participants (and the two treatment groups) will receive usual community mental healthcare services. The main services provided by the four ICCMWs mainly include day-time occupational and living skills training workshops, family mutual support groups, public and mental health education, social and recreational services, supportive groups services on specific mental health problems, referrals to community psychiatric and social care services, and individual and family counseling service as needed. In addition, the center users will also receive community mental health services provided by public hospital and outpatient departments.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: AIM_AT — The program consists of 10 weekly/biweekly, 2-hour sessions (4-months), based on the modified Kemp's model/manual of Adherence therapy and mindfulness-based psychoeducation program developed by the research team.
  Arms: Acceptance-based, insight-inducing medication adherence therapy (AIM-AT)
Behavioral: CPG — Psychoeducation group program (12-18 members/group) consists of 10 two-hour sessions, weekly/biweekly (similarly, 4-month duration) and is guided by a validated group-intervention protocol based on the research team's and McFarlane et al.'s psychoeducation programs for psychosis.
  Arms: Conventional Psychoeducation Group program (CPG)
Behavioral: TAU — Routine/Usual care only (control) group participants (and the two treatment groups) will receive usual community mental healthcare services.

SUMMARY:
This randomized controlled trial aimed to examine the effectiveness of a 10-session acceptance-based, insight-inducing medication adherence therapy (AIM-AT) program for recent-onset psychosis (in addition to usual care) over a 12-month follow-up (i.e., at immediate, 6-month, and 12-month post-intervention).

DETAILED DESCRIPTION:
Objectives: To evaluate the effectiveness of an Acceptance-based, Insight-inducing Medication Adherence Therapy (AIM_ AT) for recent-onset psychosis on patient outcomes over 12-month follow-up, when compared with a standardized psychoeducation group and routine care only.

Focus-group interviews will be performed on purposively selected participants to examine perceived benefits, satisfaction and limitations of the AIM_ AT.

Hypotheses: Compared with psychoeducation group and routine care only, the AIM_AT participants will indicate significantly greater improvements in patients' adherence to anti-psychotic medication and illness/treatment insight and other secondary outcomes (symptom severity, drug attitude, progress of recovery, psychosocial functioning, satisfaction with service, and re-hospitalization rate) at immediate post-intervention, and/or greater improvements in the above outcomes at 6- and 12-month follow-ups.

Design: A multi-center RCT with repeated-measures, three-arm design. Subjects: 126 Chinese patients with recent-onset psychosis ( </= 5 years) randomly selected from four Integrated Community Centers for Mental Wellness and randomly assigned into three study groups.

Instruments/outcome measures: Frequency, length of re-hospitalizations, and total number of patients being hospitalized from clinic records over 5-6 months; valid questionnaires (ARS, ITAQ, DAI, QPR, PANSS, SLOF, CSQ-8) for medication adherence, illness/treatment insight, drug attitude, recovery, symptom severity, functioning, and service satisfaction accordingly. Focus group interviews will collect views on benefits and weaknesses of the AIM_AT.

Data analysis: Comparing the mean value changes of outcomes between groups across time on intention-to-treat basis, using Mixed Modeling/GEE-test; and content analysis of data from focus-group interviews and intervention sessions will be conducted.

Expected results: The findings can provide evidence of the effectiveness of AIM_ AT for early-stage psychosis in community mental healthcare on improving patients' medication adherence, mental condition and recovery, functioning, and service satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* primarily diagnosed with psychosis (termed recent-onset), including brief, first-episode and other psychotic disorders according to the criteria of the DSM-V (American Psychiatric Association, 2013);
* had the mental illness ≤5 years (defined as recent-onset psychosis in recent literature)
* Hong Kong Chinese residents, aged 18-64 years;
* Global Assessment of Functioning scores ≥51, indicating mild to moderate symptoms and difficulties in psychosocial/occupational functioning (American Psychiatric Association, 2013), thus being mentally stable to comprehend AIM_AT and/or psychoeducation training;
* Unsatisfactory medication adherence as indicated by the Adherence Rating Scale of <2 (Hayward et al.,1995) during screening; and
* Able to read/understand Cantonese/Mandarin.

Exclusion Criteria:

* Participated in/have recently been receiving other psychotherapies;
* Having comorbidity of another mental illness (learning disability, cognitive or personality disorder) and/or clinically significant medical disease; and
* Having communication and/or visual/hearing difficulty.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence Rating Scale | Baseline (At recruitment)
  Rating (by RA and checking against patient records and center staff) on the level of medication adherence on a 5-point Likert-scale (1-'total non-adherence'; 2-' poor adherence'; 3-'inadequate adherence'; 4-'fair adherence'; and 5-'good adherence') with excellent inter-rater reliability and content validity.
Adherence Rating Scale | At immediate (1-2 weeks) post-intervention
  Rating (by RA and checking against patient records and center staff) on the level of medication adherence on a 5-point Likert-scale (1-'total non-adherence'; 2-' poor adherence'; 3-'inadequate adherence'; 4-'fair adherence'; and 5-'good adherence') with excellent inter-rater reliability and content validity.
Adherence Rating Scale | At 6 months post-intervention
  Rating (by RA and checking against patient records and center staff) on the level of medication adherence on a 5-point Likert-scale (1-'total non-adherence'; 2-' poor adherence'; 3-'inadequate adherence'; 4-'fair adherence'; and 5-'good adherence') with excellent inter-rater reliability and content validity.
Adherence Rating Scale | At 12 months post-intervention
  Rating (by RA and checking against patient records and center staff) on the level of medication adherence on a 5-point Likert-scale (1-'total non-adherence'; 2-' poor adherence'; 3-'inadequate adherence'; 4-'fair adherence'; and 5-'good adherence') with excellent inter-rater reliability and content validity.
Insight and Treatment Attitude Questionnaire (ITAQ) | At immediate (1-2 weeks) post-intervention
  The 10-item ITAQ was developed by McEvoy et al.(1989) to measure patients' insight and recognition of their illness and attitudes towards treatment/medication needs. Items are rated on 3-point Likert-scale (0= 'Not necessary to receive medication/treatment' to 2= 'Medication/treatment continued/required regularly')
Insight and Treatment Attitude Questionnaire (ITAQ) | At 6 months post-intervention
  The 10-item ITAQ was developed by McEvoy et al.(1989) to measure patients' insight and recognition of their illness and attitudes towards treatment/medication needs. Items are rated on 3-point Likert-scale (0= 'Not necessary to receive medication/treatment' to 2= 'Medication/treatment continued/required regularly')
Insight and Treatment Attitude Questionnaire (ITAQ) | At 12 months post-intervention
  The 10-item ITAQ was developed by McEvoy et al.(1989) to measure patients' insight and recognition of their illness and attitudes towards treatment/medication needs. Items are rated on 3-point Likert-scale (0= 'Not necessary to receive medication/treatment' to 2= 'Medication/treatment continued/required regularly')

SECONDARY OUTCOMES:
Drug Attitude Inventory (DAI) | At immediate post-intervention
  The DAI is a 10-item self-report scale measuring one's attitude towards drug adherence (equally balanced for True/False items) and containing two subscales (subjective positive and subjective negative attitude).
Drug Attitude Inventory (DAI) | At 6 months post-intervention
  The DAI is a 10-item self-report scale measuring one's attitude towards drug adherence (equally balanced for True/False items) and containing two subscales (subjective positive and subjective negative attitude).
Drug Attitude Inventory (DAI) | At 12 months post-intervention
  The DAI is a 10-item self-report scale measuring one's attitude towards drug adherence (equally balanced for True/False items) and containing two subscales (subjective positive and subjective negative attitude).
Frequency and length/duration of re-hospitalizations | At immediate post-intervention
  Frequency and length/duration of re-hospitalizations over past 5-6 months will be reported by participants at baseline and post-tests, and checked with their center records.
Frequency and length/duration of re-hospitalizations | At 6 months post-intervention
  Frequency and length/duration of re-hospitalizations over past 5-6 months will be reported by participants at baseline and post-tests, and checked with their center records.
Frequency and length/duration of re-hospitalizations | At 12 months post-intervention
  Frequency and length/duration of re-hospitalizations over past 5-6 months will be reported by participants at baseline and post-tests, and checked with their center records.
Questionnaire about the Process of Recovery (QPR) | At immediate post-intervention
  The QPR (Chinese version) consists of 22 items and 3 subscales (Self-empowerment [10-items]; Effective interpersonal relationships [6-items]; Rebuilding life [6-items]), rating on a 5-point Likert-scale ('0= disagree strongly' to '4= agree strongly').
Questionnaire about the Process of Recovery (QPR) | At 6 months post-intervention
  The QPR (Chinese version) consists of 22 items and 3 subscales (Self-empowerment [10-items]; Effective interpersonal relationships [6-items]; Rebuilding life [6-items]), rating on a 5-point Likert-scale ('0= disagree strongly' to '4= agree strongly').
Questionnaire about the Process of Recovery (QPR) | At 12 months post-intervention
  The QPR (Chinese version) consists of 22 items and 3 subscales (Self-empowerment [10-items]; Effective interpersonal relationships [6-items]; Rebuilding life [6-items]), rating on a 5-point Likert-scale ('0= disagree strongly' to '4= agree strongly').
Positive and Negative Syndrome Scale (PANSS) | At immediate post-intervention
  Mental state/Symptom severity is assessed with the 30-item PANSS(Kay 1987) across three subscales (positive symptoms, negative symptoms and general psychopathology). The scale is rated on a 7-point Likert-scale (1-'absent' to 7-'extreme'), for symptom severity.
Positive and Negative Syndrome Scale (PANSS) | At 6 months post-intervention
  Mental state/Symptom severity is assessed with the 30-item PANSS(Kay 1987) across three subscales (positive symptoms, negative symptoms and general psychopathology). The scale is rated on a 7-point Likert-scale (1-'absent' to 7-'extreme'), for symptom severity.
Positive and Negative Syndrome Scale (PANSS) | At 12 months post-intervention
  Mental state/Symptom severity is assessed with the 30-item PANSS(Kay 1987) across three subscales (positive symptoms, negative symptoms and general psychopathology). The scale is rated on a 7-point Likert-scale (1-'absent' to 7-'extreme'), for symptom severity.
Specific Level of Functioning Scale (SLOF) | At immediate post-intervention
  Patient functioning is measured by the 43-item SLOF (Schneider and Struening, 1983) in terms of three domains: physical functioning/personal care (12 items), social functioning (14 items) and community living skills (17 items) of psychosis sufferers, on 5-point Likert-scales.
Specific Level of Functioning Scale (SLOF) | At 6 months post-intervention
  Patient functioning is measured by the 43-item SLOF (Schneider and Struening, 1983) in terms of three domains: physical functioning/personal care (12 items), social functioning (14 items) and community living skills (17 items) of psychosis sufferers, on 5-point Likert-scales.
Specific Level of Functioning Scale (SLOF) | At 12 months post-intervention
  Patient functioning is measured by the 43-item SLOF (Schneider and Struening, 1983) in terms of three domains: physical functioning/personal care (12 items), social functioning (14 items) and community living skills (17 items) of psychosis sufferers, on 5-point Likert-scales.
Eight-item Client Satisfaction Questionnaire (CSQ-8) | At immediate post-intervention
  The CSQ-8 is well-accepted valid questionnaire to evaluate service users' opinions/conclusions about services received/receiving. Items are rated on 4-point Likert-scale (1- 'very dissatisfied' to 4- 'very satisfied').
Eight-item Client Satisfaction Questionnaire (CSQ-8) | At 6 months post-intervention
  The CSQ-8 is well-accepted valid questionnaire to evaluate service users' opinions/conclusions about services received/receiving. Items are rated on 4-point Likert-scale (1- 'very dissatisfied' to 4- 'very satisfied').
Eight-item Client Satisfaction Questionnaire (CSQ-8) | At 12 months post-intervention
  The CSQ-8 is well-accepted valid questionnaire to evaluate service users' opinions/conclusions about services received/receiving. Items are rated on 4-point Likert-scale (1- 'very dissatisfied' to 4- 'very satisfied').

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Integrated Community Centers for Mental Wellness, Hong Kong, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The names and emails of researchers can be shared openly for communication and collaboration.

REFERENCES:
- [Background] Chien WT, Mui J, Gray R, Cheung E. Adherence therapy versus routine psychiatric care for people with schizophrenia spectrum disorders: a randomised controlled trial. BMC Psychiatry. 2016 Feb 25;16:42. doi: 10.1186/s12888-016-0744-6. PMID 26911397
- [Background] Chien WT, Cheng HY, McMaster TW, Yip ALK, Wong JCL. Effectiveness of a mindfulness-based psychoeducation group programme for early-stage schizophrenia: An 18-month randomised controlled trial. Schizophr Res. 2019 Oct;212:140-149. doi: 10.1016/j.schres.2019.07.053. Epub 2019 Aug 12. PMID 31416744